CLINICAL TRIAL: NCT03538210
Title: Cohorte Obésité Bichat LOuis Mourier
Brief Title: Obesity Cohort Bichat Louis Mourier
Acronym: COBILOM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017SLX1085
Record Dates: First submitted 2018-03-06; First posted 2018-05-29 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Severe Obesity; Bariatric Surgery; Surgical Failure
Keywords: obesity, bariatric surgery, gastrointestinal functions, adipose tissu, steatohepatitis
MeSH Terms: conditions — Obesity, Morbid; Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity prevalence rapidly increased in the past decades in French population with multiple health consequences responsible for excess mortality. In the same period of time, the number of bariatric procedures have developed exponentially. Despite its great efficacy on weight loss but also on resolution of comorbidities, bariatric surgery is not without risks. Our hypothesis is that a better understanding of the physio-pathological consequences of obesity and bariatric surgery, notably on the gastrointestinal tract, may allow to improve the treatment of obesity and to find alternatives to bariatric surgery.

The main objective of this cohort study is to systematize the collection and the conservation of biological samples (blood, stomach, liver, intestine, adipose tissue) obtained during bariatric surgery, in obese subjects undergoing surgery (including sleeve gastrectomy, Roux-en-Y gastric bypass, or revisional intervention for complication or weight regain) in the University Hospital group of Paris Nord Val de Seine (HYPNVS).

The main projects that will build on this cohort will cover the physiopathology of obesity and its consequences, notably in the field of gastrointestinal tract including: modification of gastro-intestinal plasticity in severe obesity and after bariatric surgery and alterations of absorption of nutriments (lipids, proteins, carbohydrates) induced by obesity and bariatric surgery. The inclusion in this project of obese subjects before surgery, or lean or obese subjects after surgery will allow to distinguish the impact of weight loss and surgery on gastrointestinal remodeling. This cohort will also allow to characterize stomach and intestinal proteome in severe obesity and to precise the influence of tissue inflammation on metabolic disorders associated with obesity.

DETAILED DESCRIPTION:
The prevalence of obesity rapidly increased in the past decades in the French population with multiple health consequences (including hypertension, diabetes, sleep apnea syndrome, cardiovascular events, cancers…) responsible for excess mortality. In the same period of time, the number of bariatric procedures has developed exponentially. Indeed, there is presently little or no therapeutic alternatives in severe obesity, the pharmacotherapy of obesity having a poor efficacy. Despite its great efficacy on weight loss and resolution of comorbidities, bariatric surgery is not without risks. Indeed, it can be accompanied by side effects, including gastrointestinal disorders (transit disturbances, gastro-esophageal reflux, or dumping syndrome), surgical complications (gastric fistulas and bowel obstruction) and multiples nutritional deficiencies deleterious for health (anemia, neurological complication, bone loss, and protein malnutrition).

The mechanisms of development of obesity are still imperfectly known and, moreover, the observations made in murine models are not always transposable to humans. This is why it is necessary to establish human cohorts to specify better the pathophysiological mechanisms underlying the development of obesity and its complications and to identify new markers of response to medical and surgical treatments of obesity, in order to propose targeted therapies. In particular, the digestive tract, at the interface between the intake of nutrients and their metabolism, has a central role both in the development of obesity and in the effects of bariatric surgery.

Since 2000, bariatric surgery has been developed in University Hospital group of Paris Nord Val de Seine (HYPNVS) with a significant activity of about 600 procedures per year (mainly gastric bypass and sleeve gastrectomy). The well-systematized multidisciplinary clinical management makes it possible to phenotype the patients precisely. The collaboration between the obesity center and the INSERM 1149 research team promotes the implementation of transversal projects ranging from clinical research to basic research to deepen the physio-pathological mechanisms of obesity. Some perioperative biological samples (blood, DNA, adipose tissue, liver, intestine) were temporally collected in the surgical cohort of HUPNVS, leading to several research projects and international publications.

The team focuses on the mechanisms of gastrointestinal changes during obesity and bariatric surgery and previously showed profound changes in intestinal architecture, permeability, transport functions, metabolism, or in neuro-hormonal activity of the digestive tract. In these studies, it has been observed a plasticity of the epithelial cells constituting the gastrointestinal tract (including endocrine cells and enterocytes) that needs to be further documented. This plasticity that affects self-renewal, endocrine and digestive system and enteric nervous system, may allow epithelia to adapt to changes in the luminal environment (nutritional changes, modification of the microbiota, etc.) induced by obesity and bariatric surgery. Similarly, the connections of gastrointestinal tract with other tissues involved in metabolism and in particular the liver and adipose tissues affected by chronic inflammation and whose functions are impaired during obesity should be explored.

Our hypothesis is that a better understanding of the physio-pathological consequences of obesity and bariatric surgery, notably on the gastrointestinal tract, may allow to improve the treatment of obesity and to find alternatives to bariatric surgery.

The constitution of this cohort will allow to relate clinical data and biological data obtained in different organs (for example, to study the link between weight loss or nutritional status and gastrointestinal plasticity and transport functions). The collection of the samples either during the first surgery, or during surgical revision in subjects still obese (weight loss failure) or who have lost weight (cholecystectomies, gastro-esophageal reflux ...) will make it possible to study the consequences of obesity, weight loss but also of bariatric surgery independently of weight loss. In addition, the involvement of different teams with different fields of expertise will allow to compare the data obtained by different approaches and in different organs and thus advance in the inter-organ communication underlying the pathophysiology of obesity (for example, to study the link between inflammation of adipose tissue, NASH and metabolic complications of obesity). The characterization of specific markers, notably by studying the gastric and intestinal proteome of morbidly obese subjects, may make it possible to identify populations that are more at risk of developing certain complications and to open avenues for targeted therapies according to the profile of the patients. Moreover, a better understanding of the mechanisms and the digestive impact of bariatric surgery, will help to find non-surgical therapeutic alternatives.

The main objective of this cohort study is thus to systematize the collection and the conservation of biological samples (blood, stomach, liver, intestine, adipose tissue) obtained during bariatric surgery, in obese subjects undergoing surgery (including sleeve gastrectomy, Roux-en-Y gastric bypass, or revisional intervention for complication (cholecystectomies, intractable gastro-esophageal reflux...) or weight regain in HUPNVS

The main projects that will rely on the data of this cohort relates thus to: the gastrointestinal plasticity in morbid obesity; the status of nutrient absorption and metabolism in morbid obesity and the impact of bariatric surgery; the characterization of the gastric and intestinal proteome in morbid obese subjects; the link between tissue inflammation (adipose tissue, liver) and metabolic disorders.

The inclusion will be carried out the day before the intervention. The informed consent will be collected by the nutritionist or surgeon, and the clinical data will be recorded (socio-demographic and anthropometric data, comorbidities, metabolic parameters, digestive explorations). The surgery (gastric bypass, sleeve gastrectomy or revision) will be performed laparoscopically, according to usual practice. Tissue samples will be taken at the surgical site as part of usual care for liver biopsy (evaluation of NASH in this high-risk population), stomach in case of sleeve gastrectomy, or stomach and intestine in case of gastric bypass. Pieces (about 1 cm3) will be kept for research, but the samples will not be larger than those made for usual care. Blood samples (4 samples of 7 ml) and adipose tissue samples (2 aliquots of 10-15 g) at both subcutaneous (cutaneous incisions for the trocars) and visceral (large epiploon exposed during the intervention) localizations, will be collected and stored for research. They do not constitute an additional risk for the patient compared to the surgical procedure itself, apart from a minimal risk of hematoma at the site of collection. All tissue samples will be fixed and / or frozen at -80 ° C and stored in the Department of Pathology of Bichat hospital. The blood samples collected during the research will be frozen at -80 ° C and stored in a safe freezer at the center of biological resources of Bichat hospital for a period of 25 years.

The samples will then be analyzed according to the studies carried out, in the Department of Pathology for anatomo-pathological and immuno-histological studies and in INSERM unit 1149 for functional studies, generation of gastric and intestinal organoids, messenger RNA expression and biological assays, and by the other research teams for inflammation studies. At the end of the research, the samples may be used for subsequent analyzes not foreseen in the protocol which may prove to be interesting in the context of the pathology studied (obesity) according to the evolution of scientific knowledge, provided that the patient is not opposed, after being informed, as indicated in the information / consent form.

The originality of this project comes from the fact that at the moment there are very few teams in this topic that are organized to collect both precise phenotype (anthropometric data, co-morbidities) and systematic per-operative samples in patients with severe obesity. The current cohort project will allow to realize larger projects that will federate medico-surgical teams and INSERM researchers of HUPNVS. In addition, this project will facilitate interactions with other research units outside the hospital group by making available the stored samples, on topics related to obesity.

ELIGIBILITY:
Inclusion Criteria:

* severe obese subject with BMI above35 kg/m2, age above 18 ans who accept to participate
* candidate for bariatric surgery according to HAS criteria
* who will undergo either sleeve gastrectomy or gastric bypass
* or who undergoesa revisional surgery for a complication of bariatric surgery
* or who undergoes arevisional sugery fir insufficient weight loss
* covered by an health insurance

Exclusion Criteria:

* psychiatric disease or undertanding disorder
* alchool abuse or other addiction
* organ failure (including liver, heart or kidney)
* chronic life-threatening illness
* inflamatory disease or immunosuppressive treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe obese subjects operated for bariatric surgery or reoperated for complication
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
number of biological samples collected | during surgery
  liver stomach and intestin samples will be performed during surgery for usual care. Adiposes tissues and blood samples will be performed for reseach, on the surgical site

SECONDARY OUTCOMES:
modifications of gastro-intestinal plasticity induces by obesity and bariatric surgery | samples collected during surgery
  gene expression of basic helix-loop-helix transcription factors (fold increase as compared to control)
alterations of absroption and metabolism of nutriments induced by obesity and bariatric surgery | samples collected during surgery
  intestinal protein expression of monosaccharides, proteins, fatty acids and cholesterol transporters (fold increase as compare to control)
gastric and intestinal proteome | samples collected during surgery
  gastric and intestinal proteome in the obese morbid subject assessed by mass spectrometry
tissue inflammation and fibrosis | samples collected during surgery
  quantification of the inflammatory infiltrate of the visceral and subcutaneous adipose tissue, liver and intestine (number per area)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lousi Mourier (HUPNVS), Colombes, Île-de-France Region, France